CLINICAL TRIAL: NCT06945536
Title: Relation Between Insulinoresistance and Neutrophile to Lymphocyte Ratio in Post-operative Cardiac Surgery Patients.
Brief Title: Relation Between Insulinoresistance and Neutrophile to Lymphocyte Ratio in Cardiac Surgery.
Acronym: CRYSTAL
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/896
Record Dates: First submitted 2024-12-19; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2024-08

CONDITIONS: Insulin Resistance; Cardiac Surgery Requiring Cardiopulmonary Bypass; Neutrophil Lymphocyte Ratio
Keywords: post operative cardiac surgery; neutrophil and lymphocyte ratio; insulin resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients undergoing planned on-pump and off-pump cardiac surgery: Adult patients aged > 18 years undergoing planned coronary artery bypass surgery, surgical valve replacement, aortic surgery and surgery combining the listed procedures.

SUMMARY:
The University Hospital of Besançon is conducting a public interest research project called CRYSTAL, who studies the relationship between the Neutrophil to Lymphocyte ratio (NLR) and insulin resistance in post-operative cardiac surgery. This study could make it possible to determine, thanks to an easily measurable marker in the blood upon leaving the cardiac surgery operating room, which patients are at risk of developing insulin resistance and who would deserve close monitoring of glycemia following cardiac surgery.

Coronary artery bypass graft (CABG) and valve replacement surgeries under extracorporeal circulation (ECB) are considered high-risk procedures, particularly due to the inflammation generated by ECB. This inflammation is the cause of metabolic disturbances including insulin resistance, which causes stress hyperglycemia and glycemic variability that alters the prognosis. Insulin treatment is effective but requires enhanced monitoring and intensive care. Beyond discharge from intensive care, some patients still have insulin resistance that can persist for several days, and whose management cannot be optimally carried out in a conventional hospitalization department. The persistence of insulin resistance is explained by the intensity of the postoperative inflammatory reaction. The NLR is a simple and reliable indicator to quantify this inflammation.

The hypothesis of this study is therefore that the NLR could predict the onset of prolonged postoperative insulin resistance and identify patients likely to benefit from enhanced glycemic monitoring.

DETAILED DESCRIPTION:
Coronary artery bypass graft (CABG) and heart valve replacement surgeries under cardiopulmonary bypass (CPB) are considered high-risk procedures, associated with a morbidity of 14% and a mortality rate of 2-5% at 30 days.

This type of surgery provides activation of the innate and adaptive immune system that can be responsible for a systemic inflammatory response (SIRS). The significant increase in pro-inflammatory cytokines is associated with mortality in various clinical situations such as trauma, complex surgical procedures, sepsis, acute respiratory distress syndrome or cardiogenic shock. Thus, the massive activation of inflammatory mediators can be the cause of many endocrine and metabolic disturbances such as glycemia. The physiological stress caused by cardiac surgery, particularly under CPB, is responsible for the appearance of peri- and postoperative stress hyperglycemia in diabetic and non-diabetic patients. Stress hyperglycemia is observed mainly during the first 48 hours postoperatively but can persist for several days or even several weeks.

The Neutrophil to Lymphocyte ratio (NLR) is a marker that has been extensively studied for twenty years and used in various medical disciplines to assess the immune response to a stimulus, whether of infectious or non-infectious origin. This ratio reflects the dynamic relationship between innate immunity (neutrophils) and adaptive cellular immunity (lymphocytes).

The NLR has thus demonstrated its value in the stratification of mortality in major cardiac events, as a prognostic factor in different types of cancers, or as a predictor and marker of inflammation in infectious diseases and postoperative complications.

In cardiac surgery, an association between a high preoperative NLR rate and 30-day mortality is widely found in the literature. A large retrospective review of 3,027 patients showed that an NLR greater than 2.6 was an independent predictor of perioperative mortality (HR 2.15 p = 0.0001) and long-term mortality (HR 1.19, p = 0.0001). Haran et al. confirmed these results by showing that an NLR ≥ 3.23 is associated with an increase in 30-day mortality and various postoperative complications, namely an increase in postoperative creatinine, length of hospital stay in intensive care, duration of mechanical ventilation, postoperative delirium and an increased risk of return to the operating room.

Among the risk factors for postoperative complications, hyperglycemia and intra- and postoperative glycemic variability are factors that can potentially be cured by initiating insulin treatment with close monitoring of blood sugar levels, and which, if not treated, are associated with increased morbidity and mortality. Thus, during a stressful situation, there is a release of catecholamines, reactive oxygen species and pro-inflammatory cytokines, inducing a change in carbohydrate metabolism and the development of insulin resistance. This postoperative hyperglycemia is found in patients with pre-existing diabetes or not.

The duration of insulin resistance varies from one individual to another and can persist for several days. Glycemic control and administration of intravenous insulin treatment is only possible in the intensive care unit or intensive care unit to ensure the safety and effectiveness of the treatment. Indeed, glycemic control outside these sectors is difficult to achieve due to a lack of human resources and will therefore require the relay of intravenous insulin treatment by subcutaneous route. It could then be interesting to target patients at high risk of insulin resistance and persistence of this effect in order to maintain close postoperative glycemic monitoring.

The investigators therefore assume that the physiological disturbances caused by cardiac surgery include a systemic inflammatory state responsible, among other things, for a modification of the regulation of carbohydrate metabolism inducing stress hyperglycemia by insulin resistance and a modification of the interactions between neutrophils and lymphocytes inducing an increase in NLR. These two elements are themselves responsible for postoperative complications.

Immediate postoperative identification of an inflammatory state would thus make it possible to predict prolonged insulin resistance in the postoperative period of cardiac surgery and therefore to identify patients requiring close monitoring of blood glucose and therapeutic management. The investigators therefore hypothesize that the identification and quantification of the inflammatory state in the immediate postoperative period could make it possible to predict the level and duration of insulin resistance in the postoperative period of cardiac surgery. The Neutrophil to Lymphocyte ratio could be an inexpensive and easily achievable biomarker in routine practice that helps identify patients at risk of insulin resistance and therefore requiring close glucose monitoring.

EXPECTED RESULTS

In view of the studies previously conducted, the investigators expect that a patient with an increased NLR postoperatively after cardiac surgery will have greater postoperative insulin resistance and glycemic variability and will have more postoperative complications than a patient with a normal preoperative and/or postoperative NLR. This would therefore allow early identification of patients who are at greater risk of developing prolonged insulin resistance and therefore be a patient population deserving special attention in the management of postoperative stress hyperglycemia after their discharge from intensive care.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18
* Scheduled cardiac surgery
* Blood count the day of admission to the IS
* Subject not objecting to the use of their personal data and/or biological samples
* Affiliation to a French social security scheme or beneficiary of such a scheme

Exclusion Criteria:

* Immunosuppressive treatment
* Pre-existing corticosteroid therapy
* Hematological pathologies
* Current infection (current antibiotic therapy)
* Active tumor disease
* End-stage renal failure (DFG < 30 ml/min/1.73m² or on dialysis)
* Severe liver failure (TP < 50%)
* Diabetics on insulin
* Admission to a care unit other than Thoracic and Cardiovascular Surgery Intensive Care (SI CTCV) in the immediate post-operative period
* Pregnant women, parturients and breastfeeding mothers
* Persons deprived of their liberty by a judicial or administrative decision; persons subject to psychiatric care under constraint; persons admitted to a health or social establishment for purposes other than research
* Minors
* Adults subject to a legal protection measure or unable to express their consent
* Subject without health insurance
* Subject in the exclusion period of another study or provided for by the "national volunteer file"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had a cardiac surgery in CHU of Besançon
Sampling Method: Non-Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2024-08-25 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Sensibilty Insuline Index (SII) | 48 hours
  SII = Average glycemia over 24 hours (mmol/L)/Total insulin dose over 24 hours (IU/L)

SECONDARY OUTCOMES:
Insulin Dose-Response Index (IDRI) | 48 hours
  total insulin dose (IU)/ average glycemia (mmol/L)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: Undecided